CLINICAL TRIAL: NCT05108974
Title: Choline Supplementation as a Neurodevelopmental Intervention in Fetal Alcohol Spectrum Disorders Study
Acronym: CHOLINE4
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jeff Wozniak (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Jeff Wozniak, Professor, University of Minnesota
Organization: University of Minnesota (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMN-1506M74642; R01AA024123 (NIH)
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Fetal Alcohol Spectrum Disorders
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders | interventions — Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3 months choline bitartrate (Experimental): Over the 9-month study, participants will receive a total of 3 months of choline bitartrate (19 mg/kg) and a total of 6 months of placebo
  Interventions: Drug: Choline Bitartrate
- 6 months choline bitartrate (Experimental): Over the 9-month study, participants will receive a total of 6 months of choline bitartrate (19 mg/kg) and a total of 3 months of placebo
  Interventions: Drug: Choline Bitartrate

INTERVENTIONS:
Drug: Choline Bitartrate — Powdered drink mix for daily consumption
  Other Names: choline bitartrate formulated in drink mix specifically for this study

SUMMARY:
This is a randomized, double-blind controlled trial of choline supplementation in children with Fetal Alcohol Spectrum Disorders (FASD). The study is comparing two administration durations (3 months vs. 6 months) of choline. The primary outcome measures are cognitive measures.

DETAILED DESCRIPTION:
This project is the fourth in a series of randomized, double-blind controlled trials of choline bitartrate in children ages 2-5 (under 6) years with prenatal alcohol exposure. Pre-clinical data suggests that choline may attenuate the cognitive deficits caused by prenatal alcohol exposure (especially memory deficits). This study will evaluate the effects of daily choline supplementation in two dosing regimens (3 months choline vs. 6 months choline). Outcome measures include an elicited imitation memory paradigm, IQ measures, and measures of memory and executive functioning, and behavior.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2.5 years to 5 years old (<6 years of age) at enrollment
* Prenatal alcohol exposure
* Available parent or legal guardian capable of giving informed consent for participation.

Exclusion Criteria:

* History of a neurological condition (ex. epilepsy, traumatic brain injury)
* History of a medical condition known to affect brain function
* Other neurodevelopmental disorder (ex. autism, Down syndrome)
* History of very low birthweight (<1500 grams)

Ages: 30 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Elicited Imitation Memory Task (EI) (P.J. Bauer et al 1992 laboratory paradigm) | Change from baseline to 9 months
  Elicited Imitation short-delay memory measure (percent correct for recall)
Stanford-Binet Intelligence Test (SB-5) | Change from baseline to 9 months
  Stanford Binet Intelligence Test - 5th Edition
Minnesota Executive Function Scale (MEFS) | Change from baseline to 9 months
  Minnesota Executive Function Scale - Early Childhood Version
NIH Toolbox Flanker Test | Change from baseline to 9 months
  NIH Toolbox Flanker Inhibitory and Control Test
NIH Toolbox Picture Sequence Memory Test | Change from baseline to 9 months
  NIH Toolbox Picture Sequence Memory Test

SECONDARY OUTCOMES:
Child Behavior Checklist (CBCL) | Change from baseline to 9 months
  Child Behavior Checklist - Parent Report Version

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Wozniak, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No